CLINICAL TRIAL: NCT05467605
Title: Effect of Probiotics on Interleukin 6 and Transforming Growth Factor-βLevels in Critically Ill Children With Sepsis
Brief Title: Effect of Probiotics on Cytokines in Sepsis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ibrahim Abdallah, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: probiotics in pediatric sepsis
Record Dates: First submitted 2022-06-27; First posted 2022-07-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CASE, GROUP ONE (Active Comparator): Group 1 (group who will receive probiotics): one sachet contains(Lactobacillus acidophilus, lactobacillus delbruekii and lactobacillus fermentum 10 billions), dissolved in 10 ml distilled water twice a day for 7days orally or through nasogastric/orogastric tube depending on clinical status of patients.
  Interventions: Dietary Supplement: probiotics( Lactobacillus acidophilus, lactobacillus delbruekii and lactobacillus fermentum 10 billions),
- CONTROL, GROUP 2 (Placebo Comparator): GROUP 2 will receive only maltose dissolved in 10 ml of distilled water twice a day for 7 days orally or though nasogastric/orogastric tube depending on clinical status of patients.
  Interventions: Other: maltose dissolved in distilled water

INTERVENTIONS:
Dietary Supplement: probiotics( Lactobacillus acidophilus, lactobacillus delbruekii and lactobacillus fermentum 10 billions), — therapeutic intervention, Children will be randomized into two groups using sealed envelopes on admission after meeting inclusion criteria, group ONE will receive multi strain probiotic product which contains(Lactobacillus acidophilus, lactobacillus delbruekii and lactobacillus fermentum 10 billions),
  Other Names: LACTEOL FORTE
  Arms: CASE, GROUP ONE
Other: maltose dissolved in distilled water — the other group placebo (GROUP TWO ) will receive maltose dissolved in 10 ml distilled water .
  Arms: CONTROL, GROUP 2

SUMMARY:
To assess the effect of probiotics on cytokine's level(interleukin 6 and Transforming growth factor-β1)in children admitted to PICU with sepsis.

DETAILED DESCRIPTION:
Sepsis, defined as an infection with deregulated host response leading to life-threatening organ dysfunction. Historically, the term sepsis has been used to characterize life-threatening infections usually caused by bacterial pathogens if untreated progress to shock and death, It contributes to 19% of all deaths globally, with the highest age-specific incidence in children younger than 5 years of age. Pediatric sepsis resulted in 0.7% of all hospital encounters. Epidemiologic studies found an incidence of pediatric sepsis in up to 8% of all pediatric intensive care unit (PICU) admissions, contributing to 1in 4 deaths in PICUs.

Despite many advances in diagnosis and management, sepsis is associated with significant morbidity and mortality in pediatric population. The pathophysiology of systemic inflammatory response syndrome (SIRS)and sepsis is characterized by hyperactive and deregulated endogenous inflammatory mediators in a sequential manner resulting in a cytokine cascade.

Cytokines are regulators of the immune response to infection and play a key role in regulating inflammation and trauma. There are two types of cytokines. Pro-inflammatory cytokines and anti-inflammatory cytokines.

Pro-inflammatory cytokines(tumor necrosis factor [TNF]-α, interferon-γ, interleukin[IL]-1α, IL-1β, IL-6, IL-8, IL-12, IL-17) are important for initiation of an effective inflammatory response against pathogens, whereas their excess production can lead to multiple organ dysfunction syndrome (MODS) and mortality, on the other side, anti-inflammatory cytokines (IL-4, IL-10, IL-13,transforming growth factor [TGF]-β) are required for controlling and down-regulating the inflammatory response and if severe can lead to depression of the immune system.

The levels of these cytokines rise within few hours of onset of sepsis and remain elevated for days together depending on severity and duration of sepsis, baseline host factors, timing of sampling relative to onset of sepsis/septic shock, and inter-individual variation.

The gastrointestinal system seems to play a key role in the pathogenesis MODS owing to a breakdown of intestinal barrier function and increased translocation of bacteria and bacterial components into the systemic circulation.

During critical illness, alterations occur in gut micro flora owing to change in circulating stress hormones, gut ischemia, immune suppression, the use of antibiotics, and lack of nutrients due to delay in starting enteral feeding.

Probiotics are living micro-organisms that, when administered in adequate amounts, can help maintain the integrity of the intestinal barrier function by modulating the immune response. Such administration has been included in the management of critically ill patients as a therapeutic approach.

Various studies highlighted that probiotics can modulate intestinal micro biota by colonizing human GIT, preventing overgrowth of pathogens, normalizing altered intestinal flora, reducing bacterial translocation, influencing immune system, and balancing control of pro-inflammatory and anti-inflammatory Cytokines.

ELIGIBILITY:
Inclusion Criteria:

* The study will include children admitted to PICU with sepsis defined as presence of suspected or proven infection with two or more criteria for systemic inflammatory response syndrome (SIRS)

Exclusion Criteria:

* Children having contraindications to start enteral feeding.
* Children with known chronic gastrointestinal illness.
* Children known with immunodeficiency.
* Children on prior steroids or immunotherapy.

Ages: 30 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
1- To assess the effect of probiotics on cytokine levels(interleukin 6 and Transforming growth factor-β1) in probiotic group | one week
  To assess the effect of probiotics on cytokine levels(interleukin 6 and Transforming growth factor-β1) in probiotic group and To assess the change on cytokine levels (interleukin 6 and Transforming growth factor-β1) from day 1 to 7 in critically ill children with sepsis in two groups.

SECONDARY OUTCOMES:
assessment of other sepsis parameters | up to 2 weeks
  Assessment of other sepsis parameters like C-reactive protein ( CRP ) level in relation to prognosis of sepsis in the two groups.
assessment of patient general condition during pediatric intensive care admission | through admission till discharge from PICU up to one month
  The duration of ventilation, will be assessed in the two groups.
assessment of patient general condition during pediatric intensive care admission | through admission till discharge from PICU up to one month
  length of stay in the PICU, will be assessed in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: AYMAN EMIL, MD, Study Director — Professor of Pediatrics, Cairo University; HANAA RADY, MD, Study Director — Professor of Pediatrics, Cairo University
Locations (1):
- Cairo University Faculty of Medicine, Cairo, Egypt

REFERENCES:
- [Result] Angurana SK, Bansal A, Singhi S, Aggarwal R, Jayashree M, Salaria M, Mangat NK. Evaluation of Effect of Probiotics on Cytokine Levels in Critically Ill Children With Severe Sepsis: A Double-Blind, Placebo-Controlled Trial. Crit Care Med. 2018 Oct;46(10):1656-1664. doi: 10.1097/CCM.0000000000003279. PMID 29957709
- [Result] Chaudhry H, Zhou J, Zhong Y, Ali MM, McGuire F, Nagarkatti PS, Nagarkatti M. Role of cytokines as a double-edged sword in sepsis. In Vivo. 2013 Nov-Dec;27(6):669-84. PMID 24292568